CLINICAL TRIAL: NCT02442635
Title: Developing a Yoga Intervention During Cancer Chemotherapy
Brief Title: Yoga During Chemotherapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-15691; R34AT007935 (NIH); 15991 (Other: University of California, San Francisco)
Record Dates: First submitted 2015-04-30; First posted 2015-05-13 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Cancer; Sleep Disturbance; Fatigue
MeSH Terms: conditions — Neoplasms; Parasomnias; Fatigue | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Condition 1 (Experimental): Yoga Breathing
  Interventions: Behavioral: Yoga
- Condition 2 (Experimental): Static Yoga
  Interventions: Behavioral: Yoga
- Condition 3 (Experimental): Flowing Yoga
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Yoga breathing and postures; After this initial 3 arm experiment, yoga breathing and postures will be studied in combination.

SUMMARY:
This proposal aims to expand non-pharmacologic options for the control of symptoms during chemotherapy using yoga practices. It is particularly focused on sleep disturbance with a secondary focus on fatigue.

DETAILED DESCRIPTION:
Sleep disturbance is among the most common symptoms experienced by cancer patients, occurs in up to 80% of patients during chemotherapy, and results in serious impairments in quality of life. Although pharmacologic therapies improve sleep disturbance, they have numerous side effects, problems with tolerance and dependence, and are not well studied in oncology patients. While non-pharmacologic therapies may decrease sleep disturbance, the current level of evidence on their efficacy is insufficient. Fatigue occurs in up to 95% of those receiving chemotherapy, and results in major impairments in functioning and quality of life. Despite its significance, few effective treatments currently exist for fatigue. Prior studies suggest that yoga may be helpful for sleep disturbance and fatigue, but these studies have limitations. An important challenge in yoga research is that it is typically a multi-modality practice that can include physical postures, breathing practices, and/or meditation components. Prior studies have not adequately addressed the effects of individual components. Therefore, key questions remain unanswered about the most effective elements of yoga; how to best combine them for particular problems such as chemotherapy symptoms; and optimal dosing. The current study will address these gaps in the literature and perform key developmental steps to prepare for a large randomized, controlled trial (RCT). It builds on preliminary work in which yoga breathing practices during chemotherapy were found to improve sleep disturbance, showed trends toward improvements in fatigue, and were feasible to implement in patients undergoing chemotherapy. Using a mixed-methods approach to evaluate each intervention component, the investigators will pursue three closely interlinked steps in cancer patients receiving chemotherapy. In Aim 1 (n=10), the investigators will manualize an individualized approach to the yoga breathing intervention and iteratively refine it to insure feasibility and acceptability. In Aim 2 (n=20), the investigators will manualize a yoga posture intervention, evaluating both restorative/static poses and flowing poses, and perform iterative refinement to test feasibility and acceptability. In Aim 3 (n=70), the investigators will assess the final multi-modality yoga intervention to select final intervention elements and delivery methods for testing in a planned future RCT. This proposal will help to improve the treatment of debilitating cancer associated symptoms and advance approaches to developing therapeutic yoga intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Have a Karnofsky Performance Status Score of 60 or above
* Diagnosed with any cancer except acute leukemia
* Self-reported poor quality of sleep
* Receiving Chemotherapy
* Able to read, write, and understand English
* Ability to give informed consent

Exclusion Criteria:

* Diagnosed with brain metastasis
* Diagnosed with severe Chronic Obstructive Pulmonary Disease (COPD) or emphysema
* Have New York Heart Association class II or greater congestive heart failure
* Requiring chronic home oxygen therapy
* Diagnosed with a sleep disorder (e.g., sleep apnea or narcolepsy)
* Have received more than 3 prior chemotherapy regimens
* Receiving radiation therapy
* Has a less than 6 month life expectancy
* Regular yoga practice within the last 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-05; Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbance as measured by the General Sleep Disturbance Scale | 6 weeks

SECONDARY OUTCOMES:
Fatigue as measured by the Lee Fatigue Scale | 6 weeks

OTHER OUTCOMES:
Quality of Life as measured by the Multidimensional Quality of Life Scale--Cancer | 6 weeks
Depressive Symptoms as measured by the CES-D | 6 weeks
Anxiety as measured by the Spielberger State Anxiety Inventory | 6 weeks
Pain as measured by the modified Brief Pain Inventory | 6 weeks
Hot Flashes as measured by the Hot Flash Related Daily Interference Scale | 6 weeks
Mindfulness as measured by the Five Facet Mindfulness Questionnaire | 6 weeks
Body Awareness as measured by the Multidimensional Assessment of Interoceptive Awareness | 6 weeks
Coping and Self Efficacy as measured by the Coping and Self Efficacy Scale | 6 weeks
Social Support as measured by single items on social support | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anand Dhruva, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No